CLINICAL TRIAL: NCT03258931
Title: Phase III Randomized Study of Crenolanib Versus Midostaurin Administered Following Induction Chemotherapy and Consolidation Therapy in Newly Diagnosed Subjects With FLT3 Mutated Acute Myeloid Leukemia
Brief Title: Study of Crenolanib vs Midostaurin Following Induction Chemotherapy and Consolidation Therapy in Newly Diagnosed FLT3 Mutated AML
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arog Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARO-021
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Newly Diagnosed FLT3 Mutated AML
MeSH Terms: interventions — crenolanib; midostaurin; Cytarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Crenolanib (Experimental): Crenolanib following salvage chemotherapy
  Interventions: Drug: Crenolanib; Drug: Cytarabine; Drug: Duanorubicin
- Midostaurin (Active Comparator): Midostaurin following salvage chemotherapy
  Interventions: Drug: Midostaurin; Drug: Cytarabine; Drug: Duanorubicin

INTERVENTIONS:
Drug: Crenolanib — Crenolanib will be administered orally
  Other Names: Crenolanib besylate
  Arms: Crenolanib
Drug: Midostaurin — Midostaurin will be administered orally
  Arms: Midostaurin
Drug: Cytarabine — 100 mg/m² IV continuous infusion over 24 hours
Drug: Duanorubicin — 90 mg/m2 IV

SUMMARY:
A phase III randomized multi-center study designed to compare the efficacy of crenolanib with that of midostaurin when administered following induction chemotherapy, consolidation chemotherapy and bone marrow transplantation in newly diagnosed AML subjects with FLT3 mutation. About 510 subjects will be randomized in a 1:1 ratio to receive either crenolanib in addition to standard first line treatment of AML (chemotherapy and if eligible, transplantation) (arm A) or midostaurin and standard treatment (arm B). Potentially eligible subjects will be registered and tested for the presence of FLT3 mutation. Once the FLT3 mutation status is confirmed and additional eligibility is established, subject will be randomized and enter into the treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of de novo AML according to World Health Organization (WHO) 2016 classification
* Presence of FLT3-ITD and/or D835 mutation(s) in bone marrow or peripheral blood
* Age ≥ 18 years and ≤ 60 years
* Adequate hepatic function within 48 hours prior to induction chemotherapy
* Adequate renal functions within 48 hours prior to induction chemotherapy
* ECOG performance status within 48 hours prior to induction chemotherapy ≤ 3
* Eligible for intensive cytarabine/daunorubicin (7+3) chemotherapy specified

Exclusion Criteria:

* Acute promyelocytic leukemia (APL)
* Known clinically active central nervous system (CNS) leukemia
* Severe liver disease
* Active infections
* Known, active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Known infection with human immunodeficiency virus (HIV)
* Prior systemic anti-cancer treatment (e.g. chemotherapy, tyrosine kinase inhibitors, immunotherapy, or investigational agents)(except for hydroxyurea and/or leukapheresis)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 510 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 5 years

SECONDARY OUTCOMES:
Overall Survival | 7 years
Relapse free survival | 5 years
Composite complete remission rate | 5 years
Duration of response | 5 years

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - City of Hope National Medical Center, Duarte, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - US Davis Health, Sacramento, California
  - Yale Cancer Center, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Rush Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deacnss Medical Center Oncology, Boston, Massachusetts
  - Dana-Farber Cancer Insitute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - John Theurer Cancer Center at Hackensack UMC, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell PArk, Buffalo, New York
  - New York University, New York, New York
  - Mount Sinai, New York, New York
  - Columbia University, New York, New York
  - Cornell University, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - The UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Wake Forest Baptist Health, Section on Hematology & Oncology, Winston-Salem, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No